CLINICAL TRIAL: NCT04658823
Title: A Randomized Placebo-controlled Double-blind Pilot / Phase II Study to Assess the Efficacy and Safety of HOV-12020 in Patients With Cerebral Autosomal Dominant Arteriopathy With Subcortical Infarcts and Leukoencephalopathy (CADASIL)
Brief Title: Efficacy and Safety of Tocotrienols in CADASIL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hovid Berhad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T3-CAD-01
Record Dates: First submitted 2020-11-29; First posted 2020-12-09 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cadasil
Keywords: CADASIL; Tocotrienols; Vitamin E; Vascular; Stroke; Dementia; Cerebral Small Vessel Disease; Cognitive disorder; Neurovascular disease; Hereditary multi-infarct; Cerebrovascular disease
MeSH Terms: conditions — CADASIL; Stroke; Dementia; Cerebral Small Vessel Diseases; Cognitive Dysfunction; Cerebrovascular Disorders | interventions — Tocotrienols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HOV-12020 (Experimental): Palm tocotrienols complex Oral softgel capsule (containing 285mg mixed tocotrienols and tocopherol)
  Interventions: Drug: HOV-12020 (Palm tocotrienols complex)
- PLACEBO (Placebo Comparator): Placebo Oral Softgel capsule (each capsule containing vitamin E stripped soybean oil)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HOV-12020 (Palm tocotrienols complex) — Oral Softgel capsule containing mixed tocotrienols and tocopherol with enhanced absorption delivery system; 1 capsule twice daily
  Other Names: HOV-12020; Palm Vitamin E; Tocotrienols; Tocovid Suprabio
  Arms: HOV-12020
Drug: Placebo — Oral Softgel capsule containing soybean oil; 1 capsule twice daily
  Arms: PLACEBO

SUMMARY:
CADASIL is a paradigmatic cerebral small vessel disease responsible for white-matter lesions, accumulation of lacunes, microbleeds and cerebral atrophy. The disease is responsible for stroke and cognitive decline associated with motor disability. The number of incident lacunes, and amount of cerebral atrophy were recently found to have a strong relationship to cognitive decline and disability progression over 3 years in a large sample of patients. Palm tocotrienols has previously shown evidence of therapeutic effect in attenuating the progression of WMH related to sporadic cerebral small vessel disease in a randomized controlled clinical trial. We hypothesize that palm tocotrienols complex (HOV-12020) can reduce the clinical progression in CADASIL.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Participants aged 45 to 75 years inclusive, at the time of signing of informed consent
3. Confirmed Diagnosis of CADASIL, defined by either:

   * A Typical mutation in the NOTCH3 gene responsible for an odd number of cystein residue OR
   * A positive skin biopsy showing typical granular osmiophilic material (GOM) in the vascular wall of small vessels with electron microscopy
4. Presence of at least one prevalent lacune on the MRI identified on 3DT1 or FLAIR images.
5. Presence of Confluent white matter hyperintensities (WMH) on T2-weighted or FLAIR MR images (Fazekas grade 2-3).
6. MMSE score ≥15
7. mRS at 0 - 3
8. A woman of child bearing potential (WOCBP) is eligible to participate if she is not pregnant, not breastfeeding, and agrees to follow contraceptive guidance (as described in Appendix 5) provided by the study clinician during the treatment period and for 28 days after the last dose of the study treatment.
9. Capable of giving signed informed consent and have a patient representative willing to co-sign informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

1. Clinical stroke with persisting neurological deficit within 6 months prior to Screening.
2. Any other neurodegenerative disorder, such as Parkinson's disease, Alzheimer's disease, or Huntington's disease.
3. Current significant hematological, cardiac, pulmonary, metabolic, neurologic or psychiatric disorders, uncontrolled seizures, untreated hypertension, disorders increasing risk of bleeding (Hemophilia), or any other significant active medical condition which in the Investigator's opinion would impact participation in this study.
4. History of myocardial infarction within 3 months prior to Screening, or current active angina pectoris, or symptomatic heart failure.
5. History of cancer, within the past 5 years. Patients with basal cell carcinoma, squamous cell carcinoma, and Stage 1 prostate cancer can be included in the study.
6. An episode of major depression within the last 6 months prior to Screening (clinically stable minor depression is not exclusionary).
7. History of attempted suicide within 6 months prior to Screening or a positive response to items 4 or 5 of Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening and Baseline.
8. History of drug or alcohol abuse or dependence.
9. Contra-indications to MRI: presence of a pacemaker, severe claustrophobia, cochlear implants, ferromagnetic devices or clips, intracranial vascular clips, insulin pumps, metallic implants.
10. Pregnancy or breastfeeding women.
11. History of human immunodeficiency virus (HIV), hepatitis B or C.
12. History of allergy or severe intolerance to Vitamin E (tocopherols / tocotrienols).
13. Presence at Screening of alanine aminotransferase (ALT), aspartate aminotransferase (AST), amylase, or lipase 2x above the upper limit of normal (ULN) of laboratory reference range, total bilirubin 1.5x ULN, any other clinically significant laboratory abnormality.
14. Presence at Screening of Creatinine clearance <60 (estimated by Cockcroft-Gault equation).
15. Cognitive enhancers such as donepezil, are allowed only if stable dosage within 3 months prior to Screening.
16. Use of tocotrienol supplementation within 3 months prior to Screening or any current use of Vitamin E other than study drug (all other vitamin supplements are allowed, if stable dosage within 3 months prior to screening).
17. Participation in a clinical trial with investigational product (IP) within 30 days prior to Screening. Patients participating in observational studies with no IP, will be allowed to participate in this study
18. Indication for anti-coagulant therapy
19. Patients with known sensitivity to polyoxyl castor oil or risk of allergy to soybean and peanuts.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of manifestations related to clinical worsening | 24 months
  Occurrence one failure event within 24 months after Baseline. A failure event is considered when at least one of the following manifestations is detected during the study period:
  * incident stroke
  * increase of disability corresponding to an increase in the mRS score of at least 1 point to result in a score of 2 or greater
  * cognitive decline corresponding to a reduction of at least 4 points of the VADAS-Cog score

SECONDARY OUTCOMES:
Incidence of adverse events | 24 months
  Number of serious AEs, type of severe AEs, Total number of AEs

OTHER OUTCOMES:
Change of cognitive performance on CDR | 24 months
  Individual variation of different cognitive measures obtained using the Clinical Dementia Rating Scale Sum of Boxes (CDR-SB); score 0 to 18
Change of cognitive performances on MDRS | 24 months
  Individual variation of different cognitive measures obtained using the Mattis Dementia Rating Scale (MDRS); score 0 to 144
Change of cognitive performances on sub-subscale of MDRS | 24 months
  Individual variation of different cognitive measures obtained using the initiation/perseveration subscale of the MDRS (MDRS-I/P); score 0 to 37
Change of cognitive performances on TMT | 24 months
  Individual variation of different cognitive measures obtained using the Trail Making Test Part A and B time
Changes of gait and balance performances on SPPB | 24 months
  Between group difference on individual changes of the Short Physical Performance Battery (SPPB) score; score 0 (worst) to 12 (best)
Effects on Quality of life using SF3-6 | 24 months
  Between group differences in patient reported outcomes as assessed by the Short Form-36 (SF-36), score 0 to 100
Effects on Quality of life, using DAD | 24 months
  Between group differences in patient reported outcomes as assessed by the Disability Assessment for Dementia (DAD) scores; score 0 to 100

CONTACTS AND LOCATIONS:
Overall Officials: Pr Hugues Chabriat, Principal Investigator — Hôpital Lariboisière APHP; David Ho, Study Director — Hovid Berhad
Locations (1):
- Hôpital Lariboisière APHP, Paris, France

IPD SHARING:
Plan to Share IPD: No